CLINICAL TRIAL: NCT05857631
Title: Postoperative Hypofractionated Radiation in Cervical and Endometrial Tumours: Phase II Study
Acronym: PARCERII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Prachi Mittal, MD, Radiation Oncology, Assistant Professor, Tata Memorial Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3910; CTRI/2023/02/050123 (Registry Identifier: Clinical Trials Registry-India)
Record Dates: First submitted 2023-03-30; First posted 2023-05-12 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer; Endometrial Cancer
Keywords: Hypofractionated Radiation; Radiotherapy, Adjuvant; Radiotherapy, Intensity modulated; Late gastrointestinal and genitourinary toxicities
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — Radiotherapy; Cisplatin; Drug Therapy; Brachytherapy

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label phase II trial investigating the cumulative incidence of late grade ≥2 gastro-intestinal or genito-urinary toxicities in patients receiving adjuvant hypofractionated external beam radiotherapy to the pelvis for post-operative cervical or endometrial cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated Image guided External Beam Radiation (Experimental): Adjuvant hypofractionated external beam radiotherapy for post operative patients with cervical or endometrial cancer.
  Interventions: Radiation: Hypofractionated Image guided External Beam Radiation Therapy (EBRT); Drug: Cisplatin; Radiation: Vaginal brachytherapy

INTERVENTIONS:
Radiation: Hypofractionated Image guided External Beam Radiation Therapy (EBRT) — External beam radiotherapy to pelvis:
  Post operative hypofractionated external beam radiotherapy with intensity modulated/arc technique, to a dose of 39 Gy in 13 fractions, at 3 Gy per fraction, delivered once daily, 5 days a week, over 2.5-3 weeks.
  Other Names: Radiotherapy
Drug: Cisplatin — Patients who require adjuvant chemotherapy along with radiation, based on predefined risk features, will receive 5 cycles of cisplatin on a weekly basis with a dose of 40 mg/m2 by IV infusion over a period of 1 hour 2-4 hours prior to start of EBRT.
  Other Names: Chemotherapy
Radiation: Vaginal brachytherapy — Vaginal brachytherapy, two fractions of 6 Gy each, delivered 1 week apart.
  Other Names: Brachytherapy

SUMMARY:
The primary aim of the trial is to investigate the late effects of hypofractionated external radiation (39 Gy in 13 fractions) in patients requiring post-operative radiation for early-stage cervical and endometrial cancers.

DETAILED DESCRIPTION:
This is a phase II prospective study that will be accruing patients with post operative cervical or endometrial cancer requiring adjuvant pelvic radiation.

External beam radiotherapy (Intensity modulated radiotherapy/arc technique) will be delivered to pelvis to a dose of 39 Gray (Gy) in 13 fractions at 3 Gy per fraction, delivered once daily over 2.5 - 3 weeks. Treatment will be delivered with Intensity Modulated Radiotherapy (IMRT) under image guidance. Patients for whom concurrent chemotherapy is indicated (as per adverse risk features) will receive concurrent weekly cisplatin (40mg/m2) based on standard institutional protocol. All patients with post-operative cervical cancer will receive vaginal brachytherapy after the completion of external beam radiation. Patients with endometrial cancer with certain pre defined risk factors will also receive vaginal brachytherapy. The dose of vaginal brachytherapy will be 6 Gy high dose rate brachytherapy delivered as two different fractions, one week apart. Patients will be evaluated by the concerned investigators on a weekly basis during radiation therapy and all the toxicities will be documented according to the CTCAE V 5.0.

Patients will be followed up 3 monthly for the first 2 years, then 6 monthly from years 2 - 5, and annually thereafter. CTCAE version 5 will be used for toxicity grading at each follow-up. Quality of life assessment will be performed at baseline prior to the start of radiation and on follow-up at pre-specified times using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ-C30) and Cervix - 24 (CX24) for cervical cancer patients and Endometrium 24 (EN24) for endometrial cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
2. Histologically confirmed diagnosis of cervical cancer post hysterectomy with intermediate or high-risk features, requiring adjuvant EBRT ± concurrent chemotherapy OR histologically confirmed diagnosis of endometrial cancer post hysterectomy requiring adjuvant (chemo)radiotherapy to pelvis with/without vaginal brachytherapy.

Exclusion Criteria:

1. Patients with macroscopic residual disease (R+ resection) postoperatively
2. Patients requiring extended field radiotherapy (patients with involved para-aortic lymph nodes in cervical or endometrial cancer)
3. Patients treated with chemotherapy for any prior malignancy at any time
4. Patients treated with pelvic radiation previously
5. Patients with human immunodeficiency virus infection
6. Any preexisting medical conditions that may interfere with the assessment of genitourinary or gastrointestinal toxicity (This includes patients with irritable bowel syndrome, subacute intestinal obstruction, anal incontinence, hemorrhoids precluding analysis of gastro-intestinal toxicities, urinary incontinence, recurrent urinary tract infections)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2029-05-25 (Estimated); Study Completion 2029-05-25 (Estimated)

PRIMARY OUTCOMES:
3-year cumulative incidence of grade ≥2 gastrointestinal or genitourinary toxicity | Median follow up of 3 years
  To evaluate the 3-year cumulative incidence of late grade ≥2 gastrointestinal or genitourinary toxicity using CTCAE version 5 scoring receiving radiation with hypo fractionation.

SECONDARY OUTCOMES:
Pelvic Control Rate at 3 years | Median follow up of 3 years
  To report 3 year pelvic control rate (local and pelvic nodal) in patients receiving hypofractionated radiotherapy.
Disease Free Survival at 3 years | Median follow up of 3 years
  To report 3 year disease free survival in patients receiving hypo fractionated radiotherapy.
Overall Survival at 3 years | Median follow up of 3 years
  To report 3 year overall survival in patients receiving hypo fractionated radiotherapy.
Acute Toxicities Evaluation | 3 months
  Acute toxicity will be reported using CTCAE V. 5.0
Assessment of Quality of Life for cervical cancer patients | Median follow up of 3 years
  To assess quality of life in using EORTC QLQ-C30 and CX24. Quality of life will be measured using the EORTC QLQ C-30. For cervical cancer, EORTC QLQ CX24 module will be used. QOL scoring will be done as per standard recommendations outlined in EORTC QLQ C30 scoring manual. All patients will undergo QOL evaluation at baseline, after treatment and at subsequent follow-up.Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.
Assessment of Quality of Life for endometrial cancer patients | Median follow up of 3 years
  To assess quality of life in using EORTC QLQ-C30 and EN24. Quality of life will be measured using the EORTC QLQ C-30. For endometrial tumours, EORTC QLQ EN24 will be used. QOL scoring will be done as per standard recommendations outlined in EORTC QLQ C30 scoring manual. All patients will undergo QOL evaluation at baseline, after treatment and at subsequent follow-up.Scale- Not at all-1 , A little Bit-2, Quite a bit-3, very much-4.
  1 will be considered as better outcome & 4 will be considered as worst outcome.
C-MOSES scoring | Median follow up of 3 years
  To report cumulative toxicity score as assessed by C-MOSES scoring. Month and Severity Score (MOSES) will be calculated for each symptom (13 gastrointestinal and 6 genitourinary) with time weighted CTCAE toxicity, by using duration of time spent in each toxicity. Cumulative-MOSES score will be assessed for organ system (gastrointestinal and genitourinary), by summating MOSES of individual adverse event items respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prachi D Mittal, MD, Principal Investigator — Tata Memorial Hospital
Locations (2):
- India (2):
  - Advanced Centre for Treatment Research and Education in Cancer (ACTREC), Navi Mumbai, Maharahstra
  - Tata Memorial Hospital, Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No